CLINICAL TRIAL: NCT06597500
Title: A Single-Centre, Open-Label, Single Sequence Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of Single Inhaled Doses of GSK3923868 in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Itraconazole on the Concentration of GSK3923868 in the Blood in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 218376
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK3923868; Itraconazole; Pharmacokinetics; Drug interaction; Phosphatidylinositol 4-kinase beta (PI4KB)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Itraconazole

STUDY DESIGN:
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Period 1: GSK3923868 (Experimental): Participants will receive GSK3923868 on Day 1.
  Interventions: Drug: GSK3923868
- Treatment Period 2: GSK3923868 + Itraconazole (Experimental): Participants will receive itraconazole from Days 1 to 10 and GSK3923868 on Day 5.
  Interventions: Drug: GSK3923868; Drug: Itraconazole

INTERVENTIONS:
Drug: GSK3923868 — GSK3923868 will be administered.
Drug: Itraconazole — Itraconazole will be administered.
  Arms: Treatment Period 2: GSK3923868 + Itraconazole

SUMMARY:
The purpose of this study is to evaluate how itraconazole affects the blood concentration of GSK3923868 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation based on screening medical history, physical examination, vital signs, electrocardiogram (ECG) assessment, pulmonary function testing and laboratory tests.
* Body weight at least 50 kilograms (kg) and body-mass index (BMI) within the range 18.5 to 32.0 kilogram per meter squared (kg/m^2) (inclusive).
* For female participants: A female participant is eligible to participate if the participant is a woman of non-childbearing potential (WONCBP).
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) greater than (>) upper limit of normal (ULN).
* Total bilirubin > ULN (isolated bilirubin above ULN is acceptable if total bilirubin is fractionated and direct bilirubin less than (<) 35 percentage [%]).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Frederica's formula (QTcF) > 450 milliseconds (msec) at screening visit based on the average of triplicate ECGs.
* Past or intended use of over the counter or prescription medication, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) before the first dose of study treatment, unless in the opinion of the Investigator and the GSK Medical Monitor, the medication will not interfere with the study procedures or compromise participant safety.
* Recent donation of blood or blood products such that participation in this study would result in loss of blood in excess of 500 milliliters (mL) within a 56 day period.
* Exposure to more than 4 new chemical entities within 12 months before the first dosing day.
* Current enrolment or past participation in a clinical trial and has received an investigational product within the following time period before the first dosing day in this study: 30 days, 5 half lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Forced expiratory volume in 1 second (FEV1) < 80% predicted normal value.
* Presence of hepatitis B surface antigen (HBsAg) within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening.
* Positive hepatitis C ribonucleic acid (RNA) test result within 3 months prior to first dose of study intervention.
* Positive pre study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Current or history of drug abuse.
* History of regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of > 14 units for males and females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current or previous use of tobacco or nicotine containing products (e.g. cigarettes, nicotine patches or electronic devices) within 6 months before screening and/or have a smoking pack history of > 5 pack years.
* Positive breath carbon monoxide test indicative of recent smoking at screening or each in house admission to the clinical research unit.
* Sensitivity to the study interventions (GSK3923868, itraconazole or other azole antifungal agents) or components thereof, or drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Treatment Period 1: Area under plasma concentration versus time curve (AUC) from time zero to last quantifiable concentration [AUC(0-t)] for GSK3923868 without itraconazole co-administration | Up to Day 3
Treatment Period 2: AUC(0-t) for GSK3923868 with itraconazole co-administration | Up to Day 11
Treatment Period 1: AUC from time zero to infinity [AUC(0-∞)] for GSK3923868 without itraconazole co-administration | Up to Day 3
Treatment Period 2: AUC(0-∞) for GSK3923868 with itraconazole co-administration | Up to Day 11
Treatment Period 1: Maximum observed plasma concentration (Cmax) for GSK3923868 without itraconazole co-administration | Up to Day 3
Treatment Period 2: Cmax for GSK3923868 with itraconazole co-administration | Up to Day 11
Treatment Period 1: Time to Cmax (Tmax) for GSK3923868 without itraconazole co-administration | Up to Day 3
Treatment Period 2: Tmax for GSK3923868 with itraconazole co-administration | Up to Day 11

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Day 30
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of participants with serious adverse events (SAEs) | Up to Day 30
  An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is an abnormal pregnancy outcome, or is a suspected transmission of any infectious agent via an authorized medicinal product.
Number of participants with clinically significant changes in laboratory values | Up to Day 30
Number of participants with clinically significant changes in vital signs | Up to Day 30
Number of participants with clinically significant changes in 12-lead electrocardiogram (ECG) measurements | Up to Day 30
Treatment Period 2: AUC(0-t) for itraconazole and hydroxy-itraconazole | On Days 1 and 5
Treatment Period 2: AUC(0-∞) for itraconazole and hydroxy-itraconazole | On Days 1 and 5
Treatment Period 2: Cmax for itraconazole and hydroxy-itraconazole | On Days 1 and 5
Treatment Period 2: Tmax for itraconazole and hydroxy-itraconazole | On Days 1 and 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/